CLINICAL TRIAL: NCT04966715
Title: Inferior Epigastric Lymph Node (IELN) Basin as a Possible Systemic Metastatic Pathway of Colorectal Peritoneal Metastases
Brief Title: Inferior Epigastric Lymph Node in Colorectal Carcinosis
Acronym: EpiLyPath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EpiLyPath
Record Dates: First submitted 2021-06-14; First posted 2021-07-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Carcinomatosis
Keywords: Epigastric lymph node; Cytoreductive surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients planned for complete cytoreductive surgery (Experimental): Only one arm in the study. All patients operated for complete cytoreductive surgery and who signed informed consent form
  Interventions: Procedure: Epigastric lymph node biopsy

INTERVENTIONS:
Procedure: Epigastric lymph node biopsy — epigastric lymph node biopsy and analysis to evaluate rate dissemination of colorectal carcinomatosis by this way

SUMMARY:
In this study, the investigators propose to systematically collect and analyse epigastric lymph nodes during complete cytureductive surgery in patients with colorectal carcinomatosis, in order to define their role in the dissemination of colorectal metastases

DETAILED DESCRIPTION:
Colorectal cancer is a leading cause of cancer-related mortality worldwide. Twenty percent of the patients with CRC develop distant metastases. Among them, 50% have liver metastases (LM) and 25% have peritoneal metastases (PM). Half of these metastatic patients will present with liver-only hepatic metastases (HM) and a quarter will have just peritoneal metastases (PM). The peritoneum representing the second metastatic site in frequency. Patients with colorectal PM have a dismal prognosis in comparison with other metastatic sites. For patients with limited resectable peritoneal disease, surgery remains the only potentially curative option. The two major prognostic factors in patients undergoing cytoreductive surgery (CRS) for PM are the extent of the disease, as evaluated by the peritoneal cancer index (PCI) and the completeness of the resection. In patients undergoing complete macroscopic CRS, the 5-years overall survival (OS) is up to 45% in patients with a PCI <6, whereas OS falls to just 9% when PCI is >19. At the present time, however, only a minority (16%) of the patients who undergo surgery with a curative-intent for PM are cured, as indicated by disease-free survival (DFS) >10-years. Despite an aggressive combined approach (surgery and chemotherapy), most of these patients will die from loco-regional and/or systemic recurrence. This emphasizes the needs for a better characterization of the disease and for identification of more accurate selection criteria for surgery.

Very few studies have explored the pathophysiological mechanisms of PM development and progression. The main mechanism of reported peritoneal dissemination that has been reported is a stepwise dissemination including the exfoliation of tumoral cells from the primary tumour into the peritoneal cavity. The pathophysiological mechanisms underlying systemic dissemination in patients presenting with PM are also poorly understood. The most well-known lymphatic dissemination pathways from the peritoneum into supra-diaphragmatic lymph nodes (LNs) are the retroperitoneal lymphatic pathway and the cardio-phrenic LNs. The presence of involved cardio-phrenic LNs is predictive of PM involvement. However, detection of these LNs is based on imaging that has a limited sensitivity (65%) and surgical access requires the opening of the diaphragm.

Recently, the investigators reported, for the first time, a new lymphatic route of systemic dissemination of colorectal PM. The investigators reported LN metastases in the inferior epigastric LN basin (IELN). In this series, metabolic and morphologic imaging were not able to preoperatively predict the status of IELN. These LNs represent potential predictive factors of survival in patients treated for colorectal PM. The advantage of this LN basin is its easy surgical access that allows resection without increasing postoperative complications. The exact conditions for dissemination in IELN and their prognostic role remain undetermined.

The primary objective of this study is to evaluate the incidence of IELN basin involvement in patients with colorectal PM undergoing complete CRS. The secondary objectives are to evaluate the capacity of preoperative imaging to detect these lesions and to define conditions for IELN involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo complete cytoreductive surgery for peritoneal metastases from colorectal origin
* Patients with complete cytoreductive resection (R1) and a PCI< 20

Exclusion Criteria:

* Minor patients
* Patients unable to give written informed consent
* Previous surgery for colorectal cancer with iliac lymphadenectomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
to evaluate the incidence of IELN basin invasion in patients with CRPM undergoing complete CRS (CCR-0) | 2 years
  collection and analysis of IELN basin

SECONDARY OUTCOMES:
to define the risk for IELN invasion according to the mapping of PM | 2 years
  evaluation of the proportion of invaded IELN
to evaluate the predictive value of preoperative imaging for IELN invasion | 2 years
  comparison of imaged IELN and pathological analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No